CLINICAL TRIAL: NCT02419755
Title: A Phase II Study of Bortezomib and Vorinostat in Patients With Refractory or Relapsed MLL Rearranged Hematologic Malignancies
Brief Title: Bortezomib and Vorinostat in Younger Patients With Refractory or Relapsed MLL Rearranged Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual goals were no longer feasible based on restrictions imposed by the DSMB.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RELMLL; NCI-2015-00602 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Results first posted 2018-02-01 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2017-11

CONDITIONS: Mixed Lineage Acute Leukemia; Acute Myeloid Leukemia; Acute Lymphoid Leukemia
Keywords: Infant leukemia; ALL; AML; Biphenotypic leukemia; Pediatric
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Bortezomib; Vorinostat; Mitoxantrone; Cytarabine; Methotrexate; Hydrocortisone; pegaspargase; asparaginase erwinia chrysanthemi recombinant; Asparaginase; Dexamethasone; Calcium Dobesilate; Mercaptopurine; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stratum 1: Myeloid Malignancies (Experimental): Participants receive cytarabine, bortezomib, vorinostat, methotrexate, hydrocortisone, mitoxantrone as described in the Detailed Study Description.
  Interventions: Drug: Bortezomib; Drug: Vorinostat; Drug: Mitoxantrone; Drug: Cytarabine; Drug: Methotrexate; Drug: Hydrocortisone
- Stratum 2: ALL and MLM (Experimental): Participants in Stratum 2 [Acute Lymphoid Leukemia (ALL) and Mixed Lineage Malignancies (MLM)] receive mitoxantrone, PEG-L-Asparaginase (or Erwinia L-asparaginase), dexamethasone, bortezomib, vorinostat, cytarabine, methotrexate, hydrocortisone, mercaptopurine, and doxorubicin as described in the Detailed Study Description.
  Interventions: Drug: Bortezomib; Drug: Vorinostat; Drug: Mitoxantrone; Drug: Cytarabine; Drug: Methotrexate; Drug: Hydrocortisone; Drug: Peg-L-Asparaginase; Drug: Erwinia L-Asparaginase; Drug: Dexamethasone; Drug: Mercaptopurine; Drug: Doxorubicin

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be given as a 1 mg/mL solution intravenous (IV) push over 3 to 5 seconds. For subcutaneous (SQ) administration, bortezomib will be mixed at 2.5 mg/ml.
  Other Names: Velcade; PS-341; MLN341; LDP-341
Drug: Vorinostat — Vorinostat should be taken orally (PO) with food.
  Other Names: Zolinza; Suberoylanilide Hydroxamic Acid; SAHA
Drug: Mitoxantrone — Given by intravenous (IV) injection.
  Other Names: Novantrone
Drug: Cytarabine — Given by intravenous (IV) injection.
  Other Names: Ara-C; Cytosar
Drug: Methotrexate — Methotrexate will be given intrathecally (IT) along with hydrocortisone and cytarabine.
  Other Names: ITMHA; Intrathecal Triples
Drug: Hydrocortisone — Hydrocortisone will be given intrathecally (IT) along with methotrexate and cytarabine.
  Other Names: ITMHA; Intrathecal Triples
Drug: Peg-L-Asparaginase — Given by intravenous (IV) or intramuscular (IM) injection.
  Other Names: Pegaspargase; Oncaspar
  Arms: Stratum 2: ALL and MLM
Drug: Erwinia L-Asparaginase — To be used in case of allergy or intolerance to PEG-Asparaginase. Given by intravenous (IV) or intramuscular (IM) injection.
  Other Names: Erwinase
  Arms: Stratum 2: ALL and MLM
Drug: Dexamethasone — Given orally (PO) or intravenously (IV).
  Other Names: Decadron
  Arms: Stratum 2: ALL and MLM
Drug: Mercaptopurine — Given orally (PO).
  Other Names: 6-MP; Purinethol
  Arms: Stratum 2: ALL and MLM
Drug: Doxorubicin — Given intravenously (IV).
  Other Names: Adriamycin®
  Arms: Stratum 2: ALL and MLM

SUMMARY:
This study will test the safety and effectiveness of adding bortezomib and vorinostat to other chemotherapy drugs commonly used to treat relapsed or refractory leukemia. Both drugs have been approved by the Food and Drug Administration (FDA) to treat other cancers in adults, but they have not yet been approved tor treatment younger patients with leukemia.

PRIMARY OBJECTIVE

* To estimate the overall response rate of patients with MLL rearranged (MLLr) hematologic malignancies receiving bortezomib and vorinostat in combination with a chemotherapy backbone.

SECONDARY OBJECTIVES

* Estimate event-free and overall-survival.
* Describe toxicities experienced by participants during treatment.

OTHER PRESPECIFIED OBJECTIVES

* To identify all genomic lesions by comprehensive whole genome, exome and transcriptome sequencing on all patients.
* To compare minimal residual disease (MRD) results by three modalities: flow cytometry, polymerase chain reaction (PCR) and deep sequencing.

DETAILED DESCRIPTION:
All participants will undergo diagnostic lumbar puncture and intrathecal (IT) chemotherapy [Cytarabine, methotrexate, hydrocortisone (ITMHA)] prior to cycle 1. Throughout all phases of therapy, dexrazoxane will be given as supportive care for all participants prior to receiving mitoxantrone or doxorubicin.

STRATUM 1: MYELOID MALIGNANCIES:

Induction:

* Cytarabine, Days 1-5
* Bortezomib, Days 1, 4, 8, 11, 15, 18
* Vorinostat, Days 1-4, 8-11, 15-18
* ITMHA.for those with CNS1, Day 1
* ITMHA for those with CNS 2/3, Days 1, 4, 8, 11*, 15*, 18* and 22* (* Twice weekly until two negative CSF; CNS3 patients must receive at least 6 doses)
* Participants with cumulative anthracycline <460 mg/m2 also receive Mitoxantrone on Day 1
* Responders may receive up to 6 courses. ITMHA will be limited to day 1 for subsequent courses

Maintenance (bridge) therapy (1 cycle before stem cell transplant if needed)::

* Bortezomib, Days 1, 4, 8, 11, 15, 18
* Vorinostat, Days 1-4, 8-11, 15-18
* ITMHA, Day 1

STRATUM 2: Acute Lymphoid Leukemia (ALL) and Mixed Lineage Malignancies (MLL):

Induction:

* Mitoxantrone, Day 1
* PEG-L-Asparaginase (or Erwinia L-asparaginase), Day 3
* Dexamethasone, Days 1-4, 8-11, 15-18
* Bortezomib, Days 1, 4, 8, 11, 15, 18
* Vorinostat, Days 1-4, 8-11, 15-18
* ITMHA for those with CNS1, Days 1, 8, 15, and 22
* ITMHA for those with CNS2/3, Days 1, 4, 8, 11, 15, and 22
* Participants with >460 mg/m2 cumulative anthracyclines will not receive mitoxantrone

Consolidation:

* Methotrexate, Days 1 and 15
* Bortezomib, Days 8, 11, 22, 25
* Vorinostat, Days 8-11, and 22-25
* ITMHA, Days 1 and 15

Interim Maintenance:

* Mercaptopurine, Days 1-42
* Doxorubicin, Days 1 and 29
* PEG-L-asparaginase (or Erwinia L-asparaginase), Days 1, 15, and 29
* Dexamethasone, Days 8-11, 22-25, and 36-39
* Bortezomib Days 8,11,22,25,36,39
* Vorinostat, Days 8-11, 22-25, and 36-39
* ITMHA, Day 1

Reinduction:

* Mitoxantrone, Day 1
* PEG-L-asparaginase (or Erwinia L-asparaginase), Day 3
* Dexamethasone, Days 1-4, 8-11, 15-18
* Bortezomib Days 1, 4, 8, 11, 15, 18
* Vorinostat Days 1-4, 8-11, 15-18
* IT MHA Day 1

Maintenance (12 cycles):

* Mercaptopurine, Days 1-28
* Methotrexate, Days 8, 15, and 22
* Dexamethasone, Days 1-4
* Bortezomib, Days 1 and 4
* Vorinostat, Days 1-4
* ITMHA, Day 1

Bridge Therapy (1 cycle before stem cell transplant if needed):

* Bortezomib, Days 1, 4, 8, 11, 15, 18
* Vorinostat, Days 1-4, 8-11, 15-18
* Dexamethasone, Days 1-4, 8-11, 15-18
* ITMHA, Day 1

ELIGIBILITY:
INCLUSION CRITERIA:

* Age: Patient is ≤ 21 years of age (i.e., eligible until 22nd birthday).
* Diagnosis: Participant has a hematologic malignancy that is positive for MLLr as determined by fluorescent in situ hybridization (FISH) or RT-PCR, and disease meets at least one of the following criteria:

  * Relapsed after or is refractory to chemotherapy
  * Relapsed after hematopoietic stem cell transplantation (HSCT)
  * Relapsed or refractory secondary leukemia (Relapse is defined as reappearance of leukemia cells after the attainment of complete remission and refractory is defined as ≥5% blasts at the end of induction. Patients that achieved MRD negative status followed by reappearance of blasts at less than 5% are eligible.)
* Patients must have had verification of the malignancy at relapse, including immunophenotyping, to confirm diagnosis.
* Performance Level: Karnofsky ≥50% for patients >16 years of age and Lansky ≥50 for patients ≤16 years of age (See Appendix III). Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Prior therapy:

  * Patients who relapse while receiving standard ALL maintenance chemotherapy consisting of daily 6MP, weekly methotrexate, monthly vincristine, and monthly steroid pulse will not be required to have a waiting period before entry onto this study.
  * Patients who relapse on therapy other than standard ALL maintenance therapy must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
  * Cytotoxic therapy: At least 14 days since the completion of cytotoxic therapy with the exception of hydroxyurea, low dose cytarabine, and intrathecal chemotherapy which is permitted up to 24 hours prior to the start of protocol therapy. For patients with aggressive disease that is in the peripheral blood and rising, this 14 day washout period may be omitted.
  * Biologic (anti-neoplastic) agent: At least 7 days since the completion of therapy with a biologic agent or donor lymphocyte infusions (DLI). For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
  * Stem cell transplant or rescue: ≥2 months must have elapsed since the time of transplant. Patients with active graft-vs-host disease (GVHD) are not eligible.
* Organ function requirements: All patients must have:

  * Adequate renal function defined as: Creatinine clearance or radioisotope GFR ≥70 mL/min/1.73 m^2, OR adequate serum creatinine based on age/gender.
  * Adequate liver function defined as: Total bilirubin ≤ ULN for age, or if total bilirubin is > ULN, direct bilirubin is ≤ 1.4 mg/dL, AND SGPT (ALT) ≤4 x ULN for age, unless elevation due to leukemic infiltration
  * Adequate cardiac function defined as: Shortening fraction of ≥27% by echocardiogram OR Ejection fraction of ≥50% by gated radionuclide study
  * Central nervous system (CNS) function defined as: Patients with seizure disorder may be enrolled if on allowed anti-convulsants and well controlled. Benzodiazepines and gabapentin are acceptable. CNS toxicity ≤ Grade 2.
  * Adequate pulmonary function defined as FVC>50% predicted OR, if unable to perform pulmonary function testing, must maintain pulse oximetry oxygen saturation >92% on room air.

EXCLUSION CRITERIA:

* Patients requiring anticonvulsants known to activate the cytochrome p450 system, in particular anticonvulsants such as phenytoin, carbamazepine, and phenobarbital, are not eligible. Benzodiazepines and gabapentin are acceptable. Please see Appendix I for a list of drugs known to be potent inducers/inhibitors of the cytochrome p450 system and Appendix II for a list of anticonvulsants based on CYP3A4/5 enzyme induction.
* ALL patients who cannot receive any asparaginase products (E. Coli, PEG-asparaginase, or Erwinia asparaginase) on this study (eg, due to prior severe pancreatitis, stroke or other toxicity) are not eligible. Patients with clinically significant prior allergies to PEG-asparaginase are eligible if Erwinia L-asparaginase can be substituted.
* Pregnancy and breast feeding: patients who are pregnant or breast-feeding are not eligible for this study as there is as yet no available information regarding human fetal or teratogenic toxicities. Negative pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective birth control method.
* Investigational drugs: Patients who are currently receiving another investigational drug are not eligible.
* Anti-cancer agents: Patients who are currently receiving other anti-cancer agents with the exception of those delineated in the eligibility criteria.
* Infection: Patients who have an uncontrolled infection are not eligible. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines are acceptable.
* Known human immunodeficiency virus (HIV) infection (pre-study testing not required).
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, study participation, follow up, or interpretation of study research.
* Patients with Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or other inherited bone marrow failure syndromes are not eligible.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja A. Gruber, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — https://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve participants were enrolled at St. Jude Children's Research Hospital between April 2015 and October 2016.
Period: Overall Study
Arm/Group | Stratum 1: Myeloid Malignancies | Stratum 2: ALL and MLM
Started | 6 | 6
Completed | 3 | 2
Not Completed | 3 | 4
Not completed — Death | 1 | 3
Not completed — Relapse | 0 | 1
Not completed — Ineligible | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Although only 3 Stratum 1 and 4 Stratum 2 participants completed the trial, there were 4 Stratum 1 participants and 6 Stratum 2 participants evaluable for the outcome measures and adverse events. Basic Characteristics are provided for the evaluable participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1: Myeloid Malignancies | Stratum 2: ALL and MLM | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.39836 (1.22932) | 4.58224 (5.33903) | 4.10869 (4.08824)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Otherwise Specified, Spanish, Hispanic, Latino | 0 | 2 | 2
  Non Spanish speaking, Non Hispanic | 4 | 3 | 7
  South or Central American | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian and White | 0 | 1 | 1
  White | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate in All Participants
Description: For the purpose of the statistical analysis of the primary objective, response is assessed at the end of first treatment block at maximum tolerated dose of vorinostat (i.e., Induction Ia or Ib for myeloid and Induction for lymphoid and mixed lineage). Any eligible patient who starts first treatment block is considered evaluable. Response of CR, CRi, PR, or PRi is considered a success; otherwise a failure, which will include the cases of No-response, as well as off- treatment or off-study before response can be assessed, except cases found ineligible after enrollment. A patient found ineligible after enrollment will be taken off study and replaced by enrolling an additional MLLr patient.
  The rate (probability) of response will be estimated by the sample proportion of patients who responded (CR, CRi, PR, PRi) to Induction, along with the 99% confidence interval and lower confidence bound. Three interim analyses will be performed to monitor the possible lack of efficacy.
Time Frame: End of first treatment block (up to 2 months)
Population: The determination of overall response rate is contingent on the determination of the maximum tolerated dose. The study was terminated before the maximum tolerated dose was determined. Therefore, response rate cannot be calculated.
Arm/Group | Stratum 1: Myeloid Malignancies | Stratum 2: ALL and MLM
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With 3 Year Event Free Survival (EFS)
Description: All eligible patients who started the treatment will be included in this analysis. Patients later found ineligible will be replaced and excluded from the estimation. In addition to death for any reason, no-response (i.e., other than CR, CRi, PR or PRi), off-treatment or off-study (except for the reason of being found ineligible), disease progression, relapse, and second malignancies will be considered as failures. The time to EFS will be set to 0 for patients who fail to respond.
  Kaplan-Meier estimates of the OS and EFS functions will be computed, along with estimates of standard errors by the method of Peto. Three-year OS and EFS rates, as well as longer term survival rates (5 year and 10 year) will be estimated with 95% confidence intervals.
Time Frame: Three years after the last enrollment
Population: All eligible patients who started the treatment at the vorinostat maximum tolerated dose will be included in this analysis. The study was terminated before the maximum tolerated dose was determined.
Arm/Group | Stratum 1: Myeloid Malignancies | Stratum 2: ALL and MLM
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With 5- Year Event Free Survival
Description: as for outcome 2
Time Frame: Five years after the last enrollment
Population: as for outcome 2
Arm/Group | Stratum 1: Myeloid Malignancies | Stratum 2: ALL and MLM
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participant With 10-year Event Free Survival
Description: as for outcome 2
Time Frame: Ten years after the last enrollment
Population: as for outcome 2
Arm/Group | Stratum 1: Myeloid Malignancies | Stratum 2: ALL and MLM
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With 3-year Overall Survival (OS)
Description: All eligible patients who started the treatment will be included in this analysis. Patients later found ineligible will be replaced and excluded from the estimation. Death for any reason is considered as a failure.
  Kaplan-Meier estimates of the OS and EFS functions will be computed, along with estimates of standard errors by the method of Peto. Three-year OS and EFS rates, as well as longer term survival rates (5 year and 10 year) will be estimated with 95% confidence intervals.
Time Frame: Three years after the last enrollment
Population: as for outcome 2
Arm/Group | Stratum 1: Myeloid Malignancies | Stratum 2: ALL and MLM
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With 5-year Overall Survival
Description: as for outcome 5
Time Frame: Five years after the last enrollment
Population: as for outcome 2
Arm/Group | Stratum 1: Myeloid Malignancies | Stratum 2: ALL and MLM
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With 10-year Overall Survival
Description: as for outcome 5
Time Frame: Ten years after the last enrollment
Population: as for outcome 2
Arm/Group | Stratum 1: Myeloid Malignancies | Stratum 2: ALL and MLM
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Relevant Toxicities Related to Therapy
Description: Events were graded using CTCAE v. 4.0. All toxicities will be monitored until the completion of therapy (up to 500 days) for patients that do not go on to bone marrow transplant. If a patient goes on to receive a bone marrow transplant, at that point, they will no longer be monitored for toxicity, as any further toxicities may be secondary to the transplant and not the study regimen.
  This outcome reports those toxicities that are that were possibly, probably or definitely related to therapy. Participants were separately monitored for frequency of grade 5 events, grade 4 sepsis, grade 4 hemorrhage, and grade 4 hepatic toxicity across all patients in the stratum. Grade 4 and 5 events that are clearly and incontrovertibly due to extraneous causes or disease progression will be excluded. Higher grade events are considered more severe than lower grade.
Time Frame: From on-therapy date up to 18 months
Population: Although only 3 Stratum 1 and 4 Stratum 2 participants completed the trial, there were 4 Stratum 1 participants and 6 Stratum 2 participants evaluable for this outcome measures.
Measure: Number; unit: events
Arm/Group | Stratum 1: Myeloid Malignancies | Stratum 2: ALL and MLM
Number analyzed (Participants) | 4 | 6
events
  Grade 5: death | 1 | 3
  Grade 4: sepsis | 0 | 2
  Grade 4: hemorrhage | 0 | 1
  Grade 4: hepatic toxicity | 0 | 0

9. Other Pre Specified Outcome: Frequency of Identified Genomic Lesions
Description: Frequencies of the identified lesions will be described by counts and proportions. An established method (Pounds et al., 2013) will be applied to identify genes and pathways frequently hit by the genomic lesions.
Time Frame: Once at enrollment
Population: The investigator is unable to identify frequency of genomic lesions. To obtain useful information, a much larger sample size is needed. Genomic sequencing is cost-prohibitive to be performed on this small sample size where there are too few samples to obtain any useful information.
Arm/Group | Stratum 1: Myeloid Malignancies | Stratum 2: ALL and MLM
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Minimal Residual Disease (MRD)
Description: MRD will be monitored until the completion of therapy (up to 500 days) for patients that do not go on to bone marrow transplant. If a patient goes on to receive a bone marrow transplant, at that point, they will no longer be monitored for minimal residual disease.
  Concordance and associations of the MRD levels across three modalities (flow cytometry, PCR, and deep sequencing) as continuous measurements will be assessed by Pearson's and Spearman's correlations and Kendall's tau; MRD levels categorized into ordinal values will be analyzed by contingency tables with or without ordered margins.
Time Frame: Various time points until completion of therapy (up to 18 months)
Population: Data was either not collected or is incomplete for each of the 10 participants, and therefore cannot be analyzed.
Arm/Group | Stratum 1: Myeloid Malignancies | Stratum 2: ALL and MLM
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from a participant's on-study date until they were taken off study, up to 8 months. Although only 3 Stratum 1 and 4 Stratum 2 participants completed the trial, there were 4 Stratum 1 participants and 6 Stratum 2 participants evaluable for adverse events.
Arm/Group | Stratum 1: Myeloid Malignancies | Stratum 2: ALL and MLM
All-Cause Mortality (participants affected / at risk) | 4/4 | 6/6
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/6
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1: Myeloid Malignancies (N=4) | Stratum 2: ALL and MLM (N=6)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1: Myeloid Malignancies (N=4) | Stratum 2: ALL and MLM (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (4) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (3) | 3 (9)
Anemia (Blood and lymphatic system disorders) | 3 (33) | 3 (23)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (8) | 3 (7)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blood bilirubin, increased (Investigations) | 1 (3) | 1 (1)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CPK increased (Investigations) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (3)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (4)
Edema, trunk (General disorders) | 0 (0) | 1 (1)
Enterocolitis, infectious (Infections and infestations) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 1 (1)
Fever (General disorders) | 2 (3) | 1 (1)
Fibrinogen, decreased (Investigations) | 0 (0) | 2 (4)
GGT, increased (Investigations) | 1 (1) | 2 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5) | 5 (19)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 4 (7)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Hypertension (Vascular disorders) | 2 (3) | 4 (8)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (2) | 3 (12)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (7) | 5 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (9) | 3 (13)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (4) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 4 (29) | 5 (26)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (8) | 5 (14)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (13)
INR increased (Investigations) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Infections and infestations, other (Infections and infestations) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (2) | 2 (4)
Lung Infection (Infections and infestations) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (14) | 3 (14)
Mucosal infection (Infections and infestations) | 1 (3) | 2 (3)
Nervous system disorders, other (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 3 (3)
Neutrophil count, decreased (Investigations) | 2 (7) | 3 (7)
General disorders (Cardiac disorders) | 1 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Periorbital infection (Infections and infestations) | 1 (2) | 0 (0)
Platelet count, decreased (Investigations) | 3 (43) | 3 (43)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 3 (3)
Serum amylase, increased (Investigations) | 0 (0) | 1 (3)
Sinus bradycardia (Cardiac disorders) | 1 (2) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1) | 3 (3)
Urinary retention (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 2 (7) | 3 (17)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early, because accrual goals were no longer feasible based on restrictions imposed by the Data Safety Monitoring Board (DSMB).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes